CLINICAL TRIAL: NCT01764828
Title: A Multi-center, Phase Ib Study of MEK (Mitogen Activated Protein Kinase/ERK Kinase) Inhibitor BAY86-9766 Plus Gemcitabine in Asian Patients With Advanced or Refractory Solid Tumors
Brief Title: BAY86-9766 Plus Gemcitabine Phase I Study in Asian
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 14747
Record Dates: First submitted 2013-01-08; First posted 2013-01-10 (Estimated); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Neoplasms
Keywords: Phase I; Pharmacokinetics; Safety measurements
MeSH Terms: conditions — Neoplasms | interventions — N-(3,4-difluoro-2-(2-fluoro-4-iodophenylamino)-6-methoxyphenyl)-1-(2,3-dihydroxypropyl)cyclopropane-1-sulfonamide; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Refametinib (BAY86-9766)+ Gemcitabine (Experimental): Single dose of BAY86-9766 on Cycle 1 Day -17; twice daily dosing every day starting on day -14, start dose 50mg bid ( 30mg or 20mg are possible based on adverse events need) in addition with Gemcitabine intravenous on day 1,8 and 15 1000mg/m2
  Interventions: Drug: Refametinib (BAY86-9766); Drug: Gemcitabine

INTERVENTIONS:
Drug: Refametinib (BAY86-9766)
Drug: Gemcitabine

SUMMARY:
This is an open-label, uncontrolled, Phase Ib study designed to evaluate the safety, tolerability, and pharmacokinetics of BAY86-9766 when given as a single agent and in combination with gemcitabine in Asian patients with advanced or refractory solid tumors.Blood samples for PK (pharmacokinetics) analyses will be collected after a single dose of BAY86-9766, multiple doses of BAY86-9766, and combination treatment of gemcitabine and BAY86-9766.

Safety evaluation will include adverse events assessment, vital signs, laboratory tests, 12-lead ECG ECG (electrocardiography), cardiac function test, and ophthalmologic examination at various time points during the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients >/= 18 years of age, with histologically or cytologically documented advanced or refractory solid tumors not amenable to standard therapy
* Patients must have at least one measurable or evaluable tumor lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
* Patients must have a life expectancy of at least 12 weeks, and an Eastern Cooperative Oncology Group Performance Status (ECOG PS) </=1.

Exclusion Criteria:

* History of cardiac disease
* Active clinically serious infections > Common Terminology Criteria for Adverse Events (CTCAE) grade 2
* Known human immunodeficiency virus (HIV) infection
* Uncontrolled seizure disorder
* Undergoing renal dialysis
* Known bleeding diathesis
* History of organ allograft
* Pregnant or breast feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-02-05 (Actual); Primary Completion 2014-12-18 (Actual); Study Completion 2015-02-10 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of BAY86-9766 | Multiple time points up to 6 day
Plasma concentration of M17 and M11 | Multiple time points up to 6 day
Plasma concentration of Gemcitabine | Multiple time points up to 6 day
Plasma concentration of dFdU | Multiple time points up to 6 day
Number of adverse events, or abnormal parameters as a measure of safety and tolerability | Up to 1 year
  Parameters are laboratory parameters, vital signs, ECG parameters, cardiac function, and parameters of ophthalmologic examinations

SECONDARY OUTCOMES:
Efficacy of BAY86-9766 shown by a discrete scale | Up to 1 year
  Elements of the scale are :Complete Response (CR), Partial Response (PR), Stable Disease (SD) or Progressive Disease (PD)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (3):
- Shanghai, China
- Kashiwa, Chiba, Japan
- Seoul, South Korea